CLINICAL TRIAL: NCT02926417
Title: Interventions for Postoperative Delirium: Biomarker-2 (IPOD-B2) Pilot Study
Brief Title: Interventions for Postoperative Delirium: Biomarker-2 (IPOD-B2)
Acronym: IPOD-B2
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-0960; A530900 (Other: UW Madison); SMPH/ANESTHESIOLOGY/ANESTHESIO (Other: UW Madison); Protocol Version 4/20/2020 (Other: UW Madison)
Record Dates: First submitted 2016-09-16; First posted 2016-10-06 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participant blood and cerebral spinal fluid samples will be collected and stored for future analysis.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: High Density-Electroencephalogram

SUMMARY:
The IPOD-B2 Study aims to understand the pathogenesis of postoperative delirium in patients undergoing major surgery. The investigators will identify then correlate soluble biomarkers in blood and cerebral spinal fluid with changes in High Density-Electroencephalogram.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>21 years old)
2. Patients scheduled for an elective open thoracoabdominal aortic aneurysm or TEVAR (thoracic endovascular aortic/aneurysm repair)
3. Requiring spinal drain for surgery that is predicted to stay in two or more days
4. Willing and able to provide informed consent

Exclusion Criteria:

1. Contraindication for spinal drain
2. Documented history of dementia
3. Unable to communicate with the research staff due to language barriers
4. Individuals who the PI determines are not appropriate for the study such as a history of appointment cancellations.
5. Pregnant or Nursing
6. Prisoners

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective open thoracoabdominal aortic aneurysm or thoracic endovascular aortic/aneurysm repair surgery.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-06; Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline and correlation between biomarker levels in CSF and HD-EEG changes | Pre-operative measure: Up to 4 weeks prior to surgery. Post-operative measure: Up to postoperative day (POD) 9

SECONDARY OUTCOMES:
Absolute changes in biomarkers in CSF and plasma in delirious and non-delirious patients between baseline and post-operative period | Pre-operative measure: Up to 4 weeks prior to surgery. Post-operative measure: Up to postoperative day (POD) 9
Correlation between biomarkers in CSF and plasma in delirious and non-delirious patients | Post-operative measure: Up to postoperative day (POD) 9
Absolute changes in activity and connectivity in HD-EEG from baseline to postoperative | Pre-operative measure: Up to 4 weeks prior to surgery. Post-operative measure: Up to postoperative day (POD) 9
Correlation of biomarkers with the incidence of spinal cord ischemia | Pre-operative measure: Up to 4 weeks prior to surgery. Post-operative measure: Up to postoperative day (POD) 9

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lennertz, MD PhD, Principal Investigator — University of Wisconsin-Madison, School of Medicine and Public Health
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Taylor J, Parker M, Casey CP, Tanabe S, Kunkel D, Rivera C, Zetterberg H, Blennow K, Pearce RA, Lennertz RC, Sanders RD. Postoperative delirium and changes in the blood-brain barrier, neuroinflammation, and cerebrospinal fluid lactate: a prospective cohort study. Br J Anaesth. 2022 Aug;129(2):219-230. doi: 10.1016/j.bja.2022.01.005. Epub 2022 Feb 8. PMID 35144802
- [Derived] Tanabe S, Parker M, Lennertz R, Pearce RA, Banks MI, Sanders RD. Reduced Electroencephalogram Complexity in Postoperative Delirium. J Gerontol A Biol Sci Med Sci. 2022 Mar 3;77(3):502-506. doi: 10.1093/gerona/glab352. PMID 34958346
- [Derived] Parker M, White M, Casey C, Kunkel D, Bo A, Blennow K, Zetterberg H, Pearce RA, Lennertz R, Sanders RD. Cohort Analysis of the Association of Delirium Severity With Cerebrospinal Fluid Amyloid-Tau-Neurodegeneration Pathologies. J Gerontol A Biol Sci Med Sci. 2022 Mar 3;77(3):494-501. doi: 10.1093/gerona/glab203. PMID 34260706
- [Derived] Ballweg T, White M, Parker M, Casey C, Bo A, Farahbakhsh Z, Kayser A, Blair A, Lindroth H, Pearce RA, Blennow K, Zetterberg H, Lennertz R, Sanders RD. Association between plasma tau and postoperative delirium incidence and severity: a prospective observational study. Br J Anaesth. 2021 Feb;126(2):458-466. doi: 10.1016/j.bja.2020.08.061. Epub 2020 Nov 20. PMID 33228978
- [Derived] Tanabe S, Mohanty R, Lindroth H, Casey C, Ballweg T, Farahbakhsh Z, Krause B, Prabhakaran V, Banks MI, Sanders RD. Cohort study into the neural correlates of postoperative delirium: the role of connectivity and slow-wave activity. Br J Anaesth. 2020 Jul;125(1):55-66. doi: 10.1016/j.bja.2020.02.027. Epub 2020 Jun 1. PMID 32499013